CLINICAL TRIAL: NCT01857284
Title: A Randomized, Double-blinded, Double-dummy, Parallel-controlled and Multicenter Clinical Trial to Investigate Safety and Efficacy of Tauroursodeoxycholic Acid Capsules in Treatment of Adult Primary Biliary Cirrhosis
Brief Title: Safety and Efficacy of Tauroursodeoxycholic Acid Versus Ursofalk in the Treatment of Adult Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Trendful Kangjian Medical Information Consulting Limited Company (Other)
Responsible Party: Principal Investigator, Jia Ji-Dong, Professor, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009L05707
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Tauroursodeoxycholic Acid; Primary Biliary Cirrhosis; Safety; Efficacy
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — ursodoxicoltaurine; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Tauroursodeoxycholic Acid Capsules,250mg,tid.
  Interventions: Drug: Tauroursodeoxycholic Acid Capsules
- Group 2 (Active Comparator): Ursodeoxycholate acid capsules, 250mg,tid,
  Interventions: Drug: Ursodeoxycholic Acid Capsules

INTERVENTIONS:
Drug: Tauroursodeoxycholic Acid Capsules — 250mg.tid.po
  Other Names: Taurolite
  Arms: Group 1
Drug: Ursodeoxycholic Acid Capsules — 250mg.tid.po
  Other Names: Ursofalk
  Arms: Group 2

SUMMARY:
Though ursodeoxycholate acid (UDCA) is the wellknown effective therapy for PBC, clinical effectiveness of UDCA may be limited by its poor absorption and extensive biotransformation. The more hydrophilic bile acid tauroursodeoxycholate (TUDCA) is the active ingredients of UDCA, and has been approved by state food and drug administration in China for treatment of cholesterol stones. So it is necessary to verify the efficacy and safety of TUDCA in the treatment of adult primary biliary cirrhosis. In this randomized, double-blinded, double-dummy, parallel-controlled and multicenter clinical trial, we detect the proportion of patients who had AKP decline more than 25% as the primary outcome; decline of AKP, total bilirubin, GGT, ALT and AST as secondary outcomes after patients were treated with TUDCA or UDCA for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* aged 18-70 years
* increase in alkaline phosphatase for 2 folds or more
* positive anti-mitochondrial antibody (AMA) with presence of antibodies against the pyruvate dehydrogenase complex (AMA-M2)；AMA-negative patients should be diagnosed as PBC with histologic evidence.

Exclusion Criteria:

1. patients who had been treated with UDCA, immunosuppressive medications within 3 months.
2. patients who had evidence of extrahepatic biliary obstruction
3. patients coinfection with HBV or HCV
4. patients with one of the followings: 1) hemoglobin(HB): <11 g/dl in male, <10 g/dl in female 2) white blood cell count <3000/mm3 3) neutrophile granulocyte <1500/mm3 4) platelet <50000/mm3; 5) serum albumin <3.3 g/dl 6) alanine aminotransferase(ALT)≥10×ULN and/or aspartate aminotransferase(ALT)≥10×ULN; 7) ALT≥5×ULN and/or AST≥5×ULN coexisting with immunoglobulin G (IgG) ≥2×ULN; 8) total bilirubin ≥4×ULN; 9) prothrombin time (PT) prolong 3 seconds or more, or PTA ≦60%; 10) creatinine ≥4×ULN.
5. patients with evidence of decompensated liver disease(ascites, gastrointestinal bleeding, hepatic encephalopathy et al.)
6. definitely diagnosed as hepatocellular carcinoma(HCC), probable HCC, AFP>100ng/ml.Patients with AFP>2×ULN while <100ng/ml should re-test 2 weeks later.
7. Body Mass Index >28 kg/m2
8. drug or alcohol abuse.
9. patient with severe disease of heart, lung, kidney, alimentary canal, neural system, autoimmune disease or tumor
10. patient had or on the scheduled of organ transplantation;
11. patient for whom the follow-up is considered impossible
12. pregnant or nursing woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who had AKP decline more than 25% after 24 weeks treatment of UDCA | 12 months

SECONDARY OUTCOMES:
ALP decline from baseline after 24 weeks treatment of TUDCA | 12 month
Total bilirubin decline from baseline after 24 weeks treatment of TUDCA | 12 months
GGT decline from baseline after 24 weeks treatment of TUDCA | 12 months
ALT and AST decline from baseline after 24 weeks treatment of TUDCA | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ji Jia, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (25):
- China (25):
  - Beijing 302 Hospital, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peiking University First Hosptial, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital,SunYat-Sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Third Affiliated Hospital,SunYat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital, Wuhan, Hunan
  - 85 Military Hospital, Shanghai, Shanghai Municipality
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - NO.3 People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - RenJi Hospital, Shanghai, Shanghai Municipality
  - RuiJin Hospital, Shanghai, Shanghai Municipality
  - ShangHai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xian, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - First Affiliated Hospital Of KunMing Medical College, Kunming, Yunnan
  - The Sixth People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - First Affiliated Hospital of Zhejiang University, Zhejiang, Zhejiang